CLINICAL TRIAL: NCT02733185
Title: Trial to Assess Chelation Therapy 2
Acronym: TACT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Duke Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Gervasio Lamas, MD, TACT2 Study Chair, Mt. Sinai Medical Center, Miami
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: AT009149-01; UH3AT009149 (NIH); UH3AT009150 (NIH); R01AT009273 (NIH); U24AT009150 (NIH)
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Results first posted 2024-10-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Diabetes; Myocardial Infarction
Keywords: chelation
MeSH Terms: conditions — Diabetes Mellitus; Myocardial Infarction | interventions — Edetic Acid; Minerals

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Active/Active (Active Comparator): Active disodium EDTA (chelation) + Active Oral Multi Vitamins/Minerals (OMVM)
  Interventions: Drug: disodium EDTA; Dietary Supplement: Oral Multi Vitamins/Minerals (OMVM)
- Active/Placebo (Active Comparator): Active disodium EDTA (chelation) + Placebo Oral Multi Vitamins/Minerals (OMVM)
  Interventions: Drug: disodium EDTA
- Placebo/ Active (Active Comparator): Placebo disodium EDTA (chelation) + Active Oral Multi Vitamins/Minerals (OMVM)
  Interventions: Dietary Supplement: Oral Multi Vitamins/Minerals (OMVM); Drug: Placebo disodium EDTA
- Placebo/Placebo (Placebo Comparator): Placebo disodium EDTA (chelation) + Placebo Oral Multi Vitamins/Minerals (OMVM)
  Interventions: Drug: Placebo disodium EDTA; Dietary Supplement: Placebo Oral Multi Vitamins/Minerals (OMVM)

INTERVENTIONS:
Drug: disodium EDTA — IV Disodium Ethylene diamine tetra acetic acid in 500 cc
  Other Names: EDTA
  Arms: Active/Active; Active/Placebo
Dietary Supplement: Oral Multi Vitamins/Minerals (OMVM) — 6 tablets of Multi-vitamin/Multimineral daily
  Arms: Active/Active; Placebo/ Active
Drug: Placebo disodium EDTA — IV Placebo comparator- 500 normal saline
  Arms: Placebo/ Active; Placebo/Placebo
Dietary Supplement: Placebo Oral Multi Vitamins/Minerals (OMVM) — 6 tablets of a placebo Multi-vitamin/Multimineral daily
  Arms: Placebo/Placebo

SUMMARY:
Trial to Assess Chelation Therapy 2 (TACT2) is a randomized, double blind controlled factorial clinical trial of edetate disodium-based chelation and high-dose oral vitamins and minerals to prevent recurrent cardiac events in diabetic patients with a prior myocardial infarction (MI).

DETAILED DESCRIPTION:
The primary objective of TACT2, therefore, is to determine if the chelation-based strategy increases the time to the first occurrence of any of the components of the TACT2 primary endpoint: all-cause mortality, myocardial infarction, stroke, coronary revascularization, or hospitalization for unstable angina compared to the placebo chelation strategy.

TACT2 is a 2x2 factorial trial testing 40-weekly edetate disodium-based chelation infusions and twice daily high-dose oral multivitamins and multiminerals (OMVM) in a placebo-controlled design.

TACT2 is being carried out to replicate the findings of TACT1, which found a striking reduction of recurrent cardiovascular events in post-MI diabetic patients receiving edetate disodium-based chelation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 50 years
2. History of diabetes, defined as medical record evidence or patient report of currently using insulin or oral hypoglycemic agents, or with a history of fasting blood glucose measurement of 126 mg/dL or higher, or a history of HbA1c of 6.5% or higher.
3. History of myocardial infarction based on the Universal Definition of MI.

   1. When information about the MI hospitalization is available, all MI types except Type 2 qualify for study entry.
   2. When information about the MI hospitalization is not available, a wall motion abnormality on imaging or a perfusion defect on scan that corresponds to a coronary distribution, whether or not accompanied by pathological Q waves in the appropriate distribution, will qualify the patient for study entry. This criterion requires a call to the CCC for case review.

Exclusion Criteria:

1. Baseline serum creatinine >2.0 mg/dL.
2. HbA1C >11%.
3. Myocardial infarction within 6 weeks of randomization.
4. History of allergic reactions to EDTA or any other components of the chelation solution, including heparin. Site personnel are to call the CCC to discuss heparin allergy.
5. Coronary or peripheral arterial revascularization procedure performed within the last 6 months.
6. Planned revascularization procedure in the 6 months following enrollment.
7. Heart failure hospitalization within 6 months prior to enrollment or in clinical heart failure at the time of proposed enrollment (such as NYHA Class 3 dyspnea + rales >basilar, and additional signs of fluid overload). Such patients may be treated with diuretics and enrolled when stable.
8. Poor or no venous access in the upper extremities.
9. a. Prior intravenous chelation therapy consisting of > 1 infusion within 5 years; if only 1 infusion took place, patient cannot be enrolled for at least 12 months after said infusion.

   b. Oral chelation therapy with an approved oral chelating agent within 2 years.
10. Prior participation in TACT.
11. Baseline platelet count <100,000.
12. History of cigarette smoking within the last 3 months.
13. ALT or AST > 2.0 times the upper limit of normal.
14. Wilson's disease, hemochromatosis, or parathyroid disease.
15. Any medical condition including a current diagnosis of cancer (except non-melanoma skin cancer) that will limit patient survival over the duration of the trial.
16. Any factor that suggests that the potential participant will not be able to adhere to the protocol.
17. Women of child-bearing potential including those with plans for post-menopausal in vitro fertilization or other reproductive technology.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gervasio A Lamas, MD, Study Chair — Mount Sinai Medical Center of Florida; Kevin J Anstrom, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Daniel B Mark, MD, Principal Investigator — Duke University (Duke Clinical Research Institute)
Locations (1):
- Mount Sinai Medical Center, Miami Beach, Florida, United States

REFERENCES:
- [Background] Lamas GA, Goertz C, Boineau R, Mark DB, Rozema T, Nahin RL, Lindblad L, Lewis EF, Drisko J, Lee KL; TACT Investigators. Effect of disodium EDTA chelation regimen on cardiovascular events in patients with previous myocardial infarction: the TACT randomized trial. JAMA. 2013 Mar 27;309(12):1241-50. doi: 10.1001/jama.2013.2107. PMID 23532240
- [Background] Escolar E, Lamas GA, Mark DB, Boineau R, Goertz C, Rosenberg Y, Nahin RL, Ouyang P, Rozema T, Magaziner A, Nahas R, Lewis EF, Lindblad L, Lee KL. The effect of an EDTA-based chelation regimen on patients with diabetes mellitus and prior myocardial infarction in the Trial to Assess Chelation Therapy (TACT). Circ Cardiovasc Qual Outcomes. 2014 Jan;7(1):15-24. doi: 10.1161/CIRCOUTCOMES.113.000663. Epub 2013 Nov 19. PMID 24254885
- [Background] Lamas GA, Boineau R, Goertz C, Mark DB, Rosenberg Y, Stylianou M, Rozema T, Nahin RL, Terry Chappell L, Lindblad L, Lewis EF, Drisko J, Lee KL. EDTA chelation therapy alone and in combination with oral high-dose multivitamins and minerals for coronary disease: The factorial group results of the Trial to Assess Chelation Therapy. Am Heart J. 2014 Jul;168(1):37-44.e5. doi: 10.1016/j.ahj.2014.02.012. Epub 2014 Apr 2. PMID 24952858
- [Background] Lamas GA, Goertz C, Boineau R, Mark DB, Rozema T, Nahin RL, Drisko JA, Lee KL. Design of the Trial to Assess Chelation Therapy (TACT). Am Heart J. 2012 Jan;163(1):7-12. doi: 10.1016/j.ahj.2011.10.002. PMID 22172430
- [Background] Lamas GA, Anstrom KJ, Navas-Acien A, Boineau R, Kim H, Rosenberg Y, Stylianou M, Jones TLZ, Joubert BR, Santella RM, Escolar E, Aude YW, Fonseca V, Elliott T, Lewis EF, Farkouh ME, Nathan DM, Mon AC, Gosnell L, Newman JD, Mark DB; TACT2 Investigators. The trial to assess chelation therapy 2 (TACT2): Rationale and design. Am Heart J. 2022 Oct;252:1-11. doi: 10.1016/j.ahj.2022.05.013. Epub 2022 May 19. PMID 35598636
- [Background] Navas-Acien A, Santella RM, Joubert BR, Huang Z, Lokhnygina Y, Ujueta F, Gurvich I, LoIacono NJ, Ravalli F, Ward CD, Jarrett JM, Salazar AL, Boineau R, Jones TLZ, Mark DB, Newman JD, Nathan DM, Anstrom KJ, Lamas GA. Baseline characteristics including blood and urine metal levels in the Trial to Assess Chelation Therapy 2 (TACT2). Am Heart J. 2024 Jul;273:72-82. doi: 10.1016/j.ahj.2024.04.005. Epub 2024 Apr 15. PMID 38621575
- [Derived] Ujueta F, Lamas GA, Anstrom KJ, Navas-Acien A, Boineau R, Rosenberg Y, Stylianou M, Jones TLZ, Joubert BR, Yu Q, Wen J, Nemeth H, Huang Z, Fonseca V, Nathan DM, Uwaifo G, Arenas IA, Luo L, Baker J, Visentin D, Paixao A, Schmedtje JF Jr, Mark DB; TACT2 Investigators. Multivitamins After Myocardial Infarction in Patients With Diabetes: A Randomized Clinical Trial. JAMA Intern Med. 2025 May 1;185(5):540-548. doi: 10.1001/jamainternmed.2024.8408. PMID 40029647
- [Derived] Lamas GA, Anstrom KJ, Navas-Acien A, Boineau R, Nemeth H, Huang Z, Wen J, Rosenberg Y, Stylianou M, Jones TLZ, Joubert BR, Yu Q, Santella RM, Mon AC, Ujueta F, Escolar E, Nathan DM, Fonseca VA, Aude YW, Ehrman JK, Elliott T, Prashad R, Lewis EF, Lopes RD, Farkouh ME, Elliott AM, Newman JD, Mark DB; TACT2 Investigators. Edetate Disodium-Based Chelation for Patients With a Previous Myocardial Infarction and Diabetes: TACT2 Randomized Clinical Trial. JAMA. 2024 Sep 10;332(10):794-803. doi: 10.1001/jama.2024.11463. PMID 39141382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1,000 patients were enrolled at 88 clinical centers from United States (83) and Canada (5). The first patient was enrolled on October 18, 2017 and the last patient on December 31, 2020. Each patient was randomly assigned to 1 of the 4 treatment groups.
Groups:
- Active/Active: Active disodium EDTA (chelation) + Active Oral Multi Vitamins/Minerals (OMVM)
  disodium EDTA
  Oral Multi Vitamins/Minerals (OMVM)
- Active/Placebo: Active disodium EDTA (chelation) + Placebo Oral Multi Vitamins/Minerals (OMVM)
  disodium EDTA
  Placebo Oral Multi Vitamins/Minerals (OMVM)
- Placebo/ Active: Placebo disodium EDTA (chelation) + Active Oral Multi Vitamins/Minerals (OMVM)
  Placebo disodium EDTA
  Oral Multi Vitamins/Minerals (OMVM)
- Placebo/Placebo: Placebo disodium EDTA (chelation) + Placebo Oral Multi Vitamins/Minerals (OMVM)
  Placebo disodium EDTA
  Placebo Oral Multi Vitamins/Minerals (OMVM)
Period: Overall Study
Arm/Group | Active/Active | Active/Placebo | Placebo/ Active | Placebo/Placebo
Started | 250 | 249 | 250 | 251
Completed | 175 | 187 | 182 | 176
Not Completed | 75 | 62 | 68 | 75
Not completed — Withdrawal by Subject | 12 | 10 | 17 | 21
Not completed — Death | 46 | 34 | 35 | 43
Not completed — Lost to Follow-up | 17 | 18 | 16 | 11

BASELINE CHARACTERISTICS:
Groups:
- Active/Placebo: Active disodium EDTA (chelation) + Placebo Oral Multi Vitamins/Minerals (OMVM)
  disodium EDTA
- Placebo/ Active: Placebo disodium EDTA (chelation) + Active Oral Multi Vitamins/Minerals (OMVM)
  Oral Multi Vitamins/Minerals (OMVM)
  Placebo disodium EDTA
- Total: Total of all reporting groups
Arm/Group | Active/Active | Active/Placebo | Placebo/ Active | Placebo/Placebo | Total
Number analyzed (Participants) | 250 | 249 | 250 | 251 | 1000
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [59 to 72] | 67 [61 to 72] | 67 [61 to 72] | 67 [61 to 72] | 67 [60 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 79 | 75 | 55 | 270
  Male | 189 | 170 | 175 | 196 | 730
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 53 | 53 | 46 | 198
  Not Hispanic or Latino | 200 | 191 | 197 | 201 | 789
  Unknown or Not Reported | 4 | 5 | 0 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 3 | 1 | 5
  Asian | 15 | 11 | 12 | 16 | 54
  Native Hawaiian or Other Pacific Islander | 5 | 3 | 5 | 5 | 18
  Black or African American | 34 | 22 | 19 | 26 | 101
  White | 186 | 194 | 204 | 194 | 778
  More than one race | 1 | 3 | 1 | 1 | 6
  Unknown or Not Reported | 9 | 15 | 6 | 8 | 38
Region of Enrollment [Number; unit: participants]
  North America | 250 | 249 | 250 | 251 | 1000
Type II Diabetes [Count of Participants; unit: Participants] | 239 | 242 | 235 | 244 | 960
Time from diabetes diagnosis to randomization [Median (Inter-Quartile Range); unit: years] | 13 [7 to 20] | 15 [8 to 21] | 15 [7 to 24] | 14 [7 to 21] | 14 [7 to 22]
Time from qualifying MI to randomization [Median (Inter-Quartile Range); unit: years] | 5 [2 to 9] | 5 [2 to 10] | 5 [2 to 11] | 5 [2 to 10] | 5 [2 to 10]
Anterior MI location [Count of Participants; unit: Participants] | 71 | 73 | 80 | 86 | 310
Prior coronary revascularization [Count of Participants; unit: Participants] — Any cardiac revascularization (CABG or PCI)
  Participants | 209 | 198 | 199 | 207 | 813
Aspirin, warfarin, or P2Y12 inhibitor [Count of Participants; unit: Participants] | 223 | 224 | 225 | 225 | 897
Statin [Count of Participants; unit: Participants] | 210 | 220 | 201 | 221 | 852
Hemoglobin A1c [Median (Inter-Quartile Range); unit: %] | 7.3 [6.5 to 8.4] | 7.1 [6.4 to 8.3] | 7.3 [6.5 to 8.2] | 7.3 [6.6 to 8.5] | 7.2 [6.5 to 8.3]
HDL [Median (Inter-Quartile Range); unit: mg/dL] | 41.0 [34.0 to 49.0] | 41.0 [33.0 to 50.0] | 42.0 [35.0 to 51.0] | 40.0 [34.0 to 48.0] | 41 [34.0 to 49.0]
LDL [Median (Inter-Quartile Range); unit: mg/dL] | 75.0 [60.0 to 103.] | 72.0 [56.0 to 93.0] | 69.0 [54.0 to 87.0] | 73.0 [54.0 to 100.0] | 73 [56.0 to 96.0]
Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] | 150.0 [103.0 to 233.0] | 134.0 [100.0 to 194.0] | 139.0 [104.0 to 201.0] | 149.0 [102.0 to 226.0] | 144.0 [102.0 to 217.0]
Lead (blood) [Median (Inter-Quartile Range); unit: mcg/L] | 9.80 [6.50 to 14.69] | 8.40 [5.93 to 13.50] | 9.50 [6.41 to 14.00] | 9.20 [6.31 to 14.00] | 9.2 [6.3 to 14.0]
Cadmium (urine) [Median (Inter-Quartile Range); unit: mcg/g] | 0.27 [0.16 to 0.50] | 0.33 [0.20 to 0.55] | 0.30 [0.18 to 0.49] | 0.28 [0.18 to 0.52] | 0.30 [0.18 to 0.52]

OUTCOME MEASURES:

1. Primary Outcome: Primary Composite Outcome
Description: Time to first event: myocardial infarction, stroke, hospitalization for unstable angina, coronary revascularization, or death from any cause
Time Frame: 48 month follow-up (median)
Measure: Count of Participants; unit: Participants
Arm/Group | Active/Active | Active/Placebo | Placebo/ Active | Placebo/Placebo
Number analyzed (Participants) | 250 | 249 | 250 | 251
Participants | 85 | 89 | 90 | 86

2. Secondary Outcome: Secondary Composite Outcome
Description: Time to first event: myocardial infarction, stroke, or death from cardiovascular causes
Time Frame: 48 month follow-up (median)
Measure: Count of Participants; unit: Participants
Arm/Group | Active/Active | Active/Placebo | Placebo/ Active | Placebo/Placebo
Number analyzed (Participants) | 250 | 249 | 250 | 251
Participants | 50 | 40 | 55 | 41

3. Secondary Outcome: Secondary Outcome
Description: Time to All-Cause mortality
Time Frame: All-Cause Mortality was assessed through study completion, up to 48 months (median)
Measure: Count of Participants; unit: Participants
Arm/Group | Active/Active | Active/Placebo | Placebo/ Active | Placebo/Placebo
Number analyzed (Participants) | 250 | 249 | 250 | 251
Participants | 50 | 36 | 40 | 49

ADVERSE EVENTS:
Time Frame: All adverse events were collected from randomization until 30 days after their final infusion, approximately 13 months All-Cause Mortality was assessed through study completion, up to 48 months
Groups:
- Active EDTA/Active Vitamins: Active disodium EDTA (chelation) + Active Oral Multi Vitamins/Minerals (OMVM)
  disodium EDTA
  Oral Multi Vitamins/Minerals (OMVM)
- Active EDTA /Placebo Vitamins: Active disodium EDTA (chelation) + Placebo Oral Multi Vitamins/Minerals (OMVM)
  disodium EDTA
  Placebo Oral Multi Vitamins/Minerals (OMVM)
- Placebo EDTA/ Active Vitamins: Placebo disodium EDTA (chelation) + Active Oral Multi Vitamins/Minerals (OMVM)
  Placebo disodium EDTA
  Oral Multi Vitamins/Minerals (OMVM)
- Placebo EDTA/Placebo Vitamins: Placebo disodium EDTA (chelation) + Placebo Oral Multi Vitamins/Minerals (OMVM)
  Placebo disodium EDTA
  Placebo Oral Multi Vitamins/Minerals (OMVM)
Arm/Group | Active EDTA/Active Vitamins | Active EDTA /Placebo Vitamins | Placebo EDTA/ Active Vitamins | Placebo EDTA/Placebo Vitamins
All-Cause Mortality (participants affected / at risk) | 50/250 | 36/249 | 40/250 | 49/251
Serious Adverse Events (participants affected / at risk) | 41/250 | 40/249 | 40/250 | 40/251
Other Adverse Events (participants affected / at risk) | 0/250 | 0/249 | 0/250 | 0/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active EDTA/Active Vitamins (N=250) | Active EDTA /Placebo Vitamins (N=249) | Placebo EDTA/ Active Vitamins (N=250) | Placebo EDTA/Placebo Vitamins (N=251)
Cardiac disorders (Cardiac disorders) | 7 (7) | 15 (19) | 11 (13) | 15 (22)
Infections and infestations (Infections and infestations) | 10 (11) | 8 (10) | 17 (18) | 14 (14)
Renal and Urinary Disorders (Renal and urinary disorders) | 6 (8) | 3 (4) | 2 (2) | 3 (3)
Nervous System Disorders (Nervous system disorders) | 6 (7) | 0 (0) | 3 (3) | 6 (6)
Gastrointestinal Disorders (Gastrointestinal disorders) | 3 (6) | 5 (6) | 2 (2) | 1 (1)
General disorders and administration site conditions (General disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (5) | 5 (5) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3) | 3 (3) | 2 (2)
Vascular disorders (Vascular disorders) | 2 (3) | 2 (3) | 1 (1) | 4 (4)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 2 (4) | 2 (2) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Primary analyses were restricted to a modified intention-to-treat. Treatment adherence was imperfect. 12% of participants were lost to follow-up or withdrew consent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT02733185/Prot_001.pdf
  • Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT02733185/SAP_002.pdf
  • Informed Consent Form (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT02733185/ICF_000.pdf